CLINICAL TRIAL: NCT03967535
Title: Connectomics in Psychiatric Classification
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201404123
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Dementia; Dementia Alzheimers; Frontotemporal Dementia; Pick's Disease With Dementia
MeSH Terms: conditions — Dementia; Alzheimer Disease; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Individuals between 45-85 years old with no diagnosis of dementia. No intervention used
  Interventions: Device: MRI Brain Imaging; Behavioral: Mental Health Assessment and Computerized Cognitive Test
- Dementia: Individuals between 45-85 years old with a diagnosis of dementia. No intervention used
  Interventions: Device: MRI Brain Imaging; Behavioral: Mental Health Assessment and Computerized Cognitive Test

INTERVENTIONS:
Device: MRI Brain Imaging — Up to two Magnetic Resonance Imaging (MRI) scan sessions will be done, altogether totaling just under 3 hours of scanning. MR scanners measure brain anatomy and activity using very strong magnets. No X-rays or radiation are involved.
Behavioral: Mental Health Assessment and Computerized Cognitive Test — Participants will be asked to complete questionnaires and will be asked questions that address a broad range of personal life experiences involving social, occupational, domestic, and other behaviors.

SUMMARY:
Washington University Early Recognition Center is conducting a research study to examine brain functional connectivity and network patterns in participants with dementia.

DETAILED DESCRIPTION:
This study extends the assessment of brain connectivity and function, being conducted in the Human Connectome Project (HCP), to psychiatrically ill populations. The HCP consortium has made significant improvements in MRI instrumentation, data acquisition, preprocessing, and analysis. These improvements are currently providing publicly available data on the structure, function, and connectivity of young adult human (age 22-35) brains at unprecedented spatial resolution, temporal resolution, and accuracy. This study will focus on individuals aged 45-85 years who have a diagnosis of dementia, or are healthy controls. Additionally, similar to the HCP, the investigator will study the effect of genetics on the patterns of brain connectivity in various psychiatric populations. DNA will be collected non-invasively from saliva. Furthermore, this investigator will study cortisol levels in hair samples as an additional assessment to help characterize brain imagining findings.

ELIGIBILITY:
Inclusion Criteria:

* Ages 45-85
* Has consented to participate or has an LAR present that has consented to participate
* DSM-5 diagnosis of Dementia

Exclusion Criteria:

* Any genetic disorder, such as cystic fibrosis or sickle cell disease
* Multiple Sclerosis
* Cerebral Palsy
* Loss of consciousness for >30 minutes
* Pregnancy
* Hospitalization for stroke, brain aneurysm, brain hemorrhage, or subdural hematoma

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 45-85 with a diagnosis of Dementia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) Brain Imaging | within one month of study enrollment
  The current project aims to uncover latent, homogenous, connectivity phenotypes using neuroimaging tools, which are free from the limitations of traditional diagnostic boundaries, and which correlate with clinical characteristics. The investigator will use resting state functional connectivity MRI (rs-fcMRI), diffusion MRI (dMRI) and tract-based spatial statistics (TBSS) to identify brain signatures that cut across psychiatric disorders.

SECONDARY OUTCOMES:
DNA testing through saliva | within one month of study enrollment
  Saliva samples will be collected from participants for DNA extraction and the development of lymphoblastoid cell lines. DNA is used for research purposes only, for studies assessing brain connectivity.

OTHER OUTCOMES:
Hair sample for cortisol measurement | within one month of study enrollment
  To see how cortisol levels can help characterize brain imaging findings

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No